CLINICAL TRIAL: NCT02621463
Title: Electric Blower Based Ventilator Used During Procedural Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kai Kuck, Ph.D., University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB_00074281
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Results first posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Apnea During Procedural Sedation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Noninvasive Ventilation (Experimental): Use of the Noninvasive Ventilator (V60, Philips). The ventilator mask will be placed on the patient's face according to their comfort using an elastomeric H-strap. CPAP of 8 cmH2O (pressure) will be the starting setting for the ventilator.
  Interventions: Device: Noninvasive Ventilator (V60, Philips)

INTERVENTIONS:
Device: Noninvasive Ventilator (V60, Philips) — The clinician will determine the concentration of oxygen that shall be delivered to the patient. The ventilator is capable of providing concentrations between 21% - 100% of oxygen. Unless otherwise directed by the clinician, the default setting of 40% will be used.

SUMMARY:
Conduct human trials in the endoscopy suite of our continuous positive airway pressure (CPAP) ventilator approach using an FDA approved ventilator.

DETAILED DESCRIPTION:
All study procedures will be performed in adult patients following informed consent at the endoscopy suite of the University of Utah Health Sciences Center in Salt Lake City, Utah. A ventilation mask will be placed on the patient's face and connected to the ventilator. Supplemental oxygen will be delivered by the ventilator through the mask; the concentration of oxygen delivered will be left to the clinician's discretion. A modified mask with multiple small leaks will be used with a standard elastomeric H-strap to secure it to the patient's face.

The endoscopy suite nurse and technicians will attach all clinically necessary standard sensors and connect them to the patient and monitoring system. Height, weight, and neck circumference will be measured and recorded digitally on an encrypted laptop. In addition to the standard of care monitors, the investigators will collect data from additional non-invasive modalities and save the data to a laptop using custom software for later analysis.

Pressure and flow sensors included in the ventilator will be used to monitor the patients' tidal volumes and respiratory rate during the procedure. The data that will be collected and recorded on the laptop will include: RIP data, mask pressure, flow, and breath rate. An additional flow sensor will be placed in line with the ventilator.

The objective of this study is threefold: Demonstrate in patients undergoing procedural sedation (e.g., for colonoscopy) that obstructive apnea can successfully be avoided by stenting the airway open using CPAP, demonstrate that we can successfully detect periods of zero ventilation, and demonstrate the functionality of the modified standard mask.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* undergoing a colonoscopy procedure
* receiving registered nurse-administered procedural sedation at the University of Utah Health Sciences Center
* agree to participate
* written informed consent

Exclusion Criteria:

* Inability/refusal of subject to provide informed consent.
* Standard colonoscopy exclusion criteria used at the GI lab at the University of Utah.
* Pregnant patients and patients with an ASA (American Society of Anesthesiology) physical status of IV or V.
* Patients with severe medical condition(s) that in the view of the acting physician prohibits participation in the study.
* Patients with a BMI > 35 will not be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kai Kuck, Ph.D., Principal Investigator — University of Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Noninvasive Ventilation
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Noninvasive Ventilation
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 29
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 27 (6)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time the Patient Will Experience Apnea
Description: Length of time in minutes the patient experiences apnea divided by the length of time of the diagnostic procedure (Unit: %)
Time Frame: Duration of Diagnostic Procedure (Colonoscopy)
Measure: Median (Inter-Quartile Range); unit: % time in apnea of total study duration
Arm/Group | Noninvasive Ventilation
Number analyzed (Participants) | 29
% time in apnea of total study duration | 11 [4 to 22]

ADVERSE EVENTS:
Time Frame: Participation and adverse event reporting was limited to the study intervention, mean of 24 minutes (SD 11).
Arm/Group | Noninvasive Ventilation
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

LIMITATIONS AND CAVEATS:
This was not a randomized clinical trial involving multiple facilities.

The pharmacodynamic effect of the sedation were unknown.

The CPAP machine and the tight-fitting mask may have provided enough of a stimulus as to maintain the patient in a lighter sedation state.

The proprietary C-flex and Auto-Trak algorithms are integrated into the V60 ventilator and could not be disabled. The algorithms did cause some variation in pressure levels delivered to the patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-30): https://cdn.clinicaltrials.gov/large-docs/63/NCT02621463/Prot_SAP_000.pdf